CLINICAL TRIAL: NCT01420445
Title: Randomized, Double-blind, Placebo/Active-controlled, Multi-center, Phase 3 Clinical Trial to Investigate the Safety/Tolerability and Efficacy of YHD001 After Oral Administration in Patients With Acute or Chronic Bronchitis
Brief Title: Safety/Tolerability and Efficacy of YHD001 in Patients With Acute and Chronic Bronchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YHD001-202
Record Dates: First submitted 2011-07-20; First posted 2011-08-19 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Acute Bronchitis; Chronic Bronchitis
MeSH Terms: conditions — Bronchitis; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- YHD001 dose level 1 (Experimental): YHD001 dose level 1
  Interventions: Drug: YHD001 dose level 1
- YHD001 dose level 2 (Experimental): YHD001 dose level 2
  Interventions: Drug: YHD001 dose level 2
- Pelargonium sidoides extract (Active Comparator): Pelargonium sidoides extract (Syrup)
  Interventions: Drug: Pelargonium sidoides extract
- Placebo (Placebo Comparator): Placebo for YHD001 & active comparator(syrup)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: YHD001 dose level 1 — three times daily / 7 days
  Other Names: Undecided
  Arms: YHD001 dose level 1
Drug: YHD001 dose level 2 — three times daily / 7 days
  Other Names: Undecided
  Arms: YHD001 dose level 2
Drug: Pelargonium sidoides extract — 6-9mL three times daily / 7 days
  Other Names: UMCKAMIN Syrup
  Arms: Pelargonium sidoides extract
Drug: placebo — three times daily / 7 days
  Arms: Placebo

SUMMARY:
The study will conduct with 4 comparative groups orally treated with YHD001 dose level 1(t.i.d.), YHD001 dose level 2(t.i.d.), pelargonium sidoides extract 9mL(t.i.d.) or Placebo for 7 days.

The treatments will be assigned randomly to patients (n=116) with acute or chronic bronchitis.

DETAILED DESCRIPTION:
The outcome measures is to evaluate the overall change from baseline to the end of treatment in scores relating to the severity of four symptom of bronchitis: cough, sputum, QOL of daily life, QOL of falling asleep at night.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥18 year
* Provision of written informed consent
* Acute bronchitis with a Bronchitis Severity Score(BSS)≥five points

Exclusion Criteria:

* History of any clinically significant disease
* History of drug/chemical/alcohol abuse
* Use of antibiotics, anti-histamine during the 7 days before administration of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of total symptom score from baseline to the end of treatment | 7 days

SECONDARY OUTCOMES:
safety assessment | 7 days
  comparison of the adverse event profiles throughout the course of the study, ECGs and safety blood tests on D0 and D7.
time to response | 7 days
compliance, defined by drug accountability | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Young Kyoon Kim, M.D., Ph.D., Principal Investigator — Division of Respiratory and Critical Care Medicine, Department of Internal Medicine, Seoul St. Mary's Hospital,College of Medicine, The Catholic University of Korea
Locations (1):
- The Catholic University of Korea Seoul St. Mary'S Hospital, Seoul, South Korea